CLINICAL TRIAL: NCT00005733
Title: Develop and Implement Asthma Controlling Strategies (2)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4942
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-09

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To develop and implement asthma controlling strategies for inner city and high risk populations.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a serious chronic disease affecting about 12 million Americans; about 3 million are children. The study was part of an initiative, "Developing and Implementing at the State and Local Level Educational Strategies and Interventions for Controlling Asthma in Inner City and High Risk Populations", released in February 1993 by the National Asthma Education Program of the Office of Prevention, Education and Control.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1997-03

REFERENCES:
- [Background] Wilson SR, Scamagas P, Grado J, Norgaard L, Starr NJ, Eaton S, Pomaville K. The Fresno Asthma Project: a model intervention to control asthma in multiethnic, low-income, inner-city communities. Health Educ Behav. 1998 Feb;25(1):79-98. doi: 10.1177/109019819802500107. PMID 9474501